CLINICAL TRIAL: NCT00788892
Title: Phase IIB, Multicenter, Randomized, Open Label Trial of CPX-351 (Cytarabine:Daunorubicin) Liposome Injection Versus Cytarabine and Daunorubicin in Patients With Untreated AML 60-75 Years of Age.
Brief Title: Trial of CPX-351 in Newly Diagnosed Elderly AML Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0308-204
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute; Myeloid; Leukemia; elderly; Newly; Diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Disease | interventions — CPX-351; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: CPX-351 (Experimental): First induction: CPX-351 at 100u/m2 administered on days 1, 3 and 5 Second induction: CPX-351 at 100u/m2 administered on days 1 and 3 Consolidation: CPX-351 at 100u/m2 administered on days 1 and 3
  Interventions: Drug: CPX-351
- Arm B: Cytarabine + Daunorubicin (Active Comparator): First induction: Cytarabine at a dose of 100mg/m2/day on days 1-7, Daunorubicin at dose of 45 or 60mg/m2 on days 1-3 Second induction: Cytarabine at a dose of 100mg/m2/day on days 1-5, Daunorubicin at a dose of 45 or 60 mg/m2/day on days 1 and 2 Consolidation: Investigator's Choice
  Interventions: Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: CPX-351
  Arms: Arm A: CPX-351
Drug: Cytarabine
  Arms: Arm B: Cytarabine + Daunorubicin
Drug: Daunorubicin
  Arms: Arm B: Cytarabine + Daunorubicin

SUMMARY:
The study investigates if CPX-351 will be a) more effective than the standard AML treatment and b) more tolerable than the standard AML treatment regimens.

The study compares the investigational product CPX-351 vs the standard treatment for AML in this patients age group.

DETAILED DESCRIPTION:
This study is a randomized, open-label, parallel-arm, fixed-dose, standard therapy controlled Phase IIB trial. Study enrollment duration is expected to be approximately 12-18 months. On entry, patients are randomized to receive either CPX-351 or standard induction treatment with cytarabine and daunorubicin("7 and 3" regimen).

Patients are stratified to balance the likelihood of obtaining a CR and the duration of CR between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 and <76 years at the time of diagnosis of AML
* Pathological confirmation of AML
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

Serum creatinine < 2.0 mg/dL Serum total bilirubin < 2.0 mg/dL Serum alanine aminotransferase or aspartate aminotransferase < 150 IU/liter Note: If elevated liver enzymes are related to disease; contact medical monitor to discuss.

* Cardiac ejection fraction > 50% by echocardiography or MUGA scan

Exclusion Criteria:

* Patients with locally advanced or metastatic solid tumors ≤5 years from initial diagnosis are excluded. (Patients with locally advanced or metastatic solid tumors >5 years from initial diagnosis, for whom the investigator has no clinical suspicion of active disease for >2 years before randomization are eligible)
* Prior treatment for AML; only hydroxyurea is permitted (see below)
* Acute promyelocytic leukemia [t(15;17)] or favorable cytogenetics, including t(8;21) or inv16 if known at the time of randomization
* Patients with a prior anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent)
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Administration of any antineoplastic therapy within 4 weeks of the first CPX-351 dose; in the event of rapidly proliferative disease use of hydroxyurea is permitted until 24 hours before the start of study treatment
* Clinical evidence of active CNS leukemia
* Patients with history of and/or current evidence of myocardial impairment (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Class III or IV staging
* Active and uncontrolled infection. Patients with an infection receiving treatment with antibiotics may be entered into the study if they are afebrile and hemodynamically stable for 72 hrs.
* Current evidence of invasive fungal infection (blood or tissue culture); HIV or active hepatitis C infection
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-related disorder

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Lancet, MD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (28):
- United States (25):
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Davis Cancer Center, Sacramento, California
  - University of California Medical Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Robert H.Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St.Francis Hospital, Beech Grove, Indiana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northern New Jersey Cancer Associates, Hackensack, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Weil Cornell Medical Center, New York, New York
  - New York Medical College, Division of Oncology, Valhalla, New York
  - Blumenthal Cancer Center/Mecklenburg Medical Group, Charlotte, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburg Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Cancer Therapy and Research Center at the University of Texas, San Antonio, Texas
  - Froedlert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - BC Cancer Research Center, Vancouver, British Columbia
  - Queen Elisabeth II Health Sciences Center, Halifax, Nova Scotia
  - McGill University Department of Oncology, Montreal, Quebec

REFERENCES:
- [Derived] Lancet JE, Cortes JE, Hogge DE, Tallman MS, Kovacsovics TJ, Damon LE, Komrokji R, Solomon SR, Kolitz JE, Cooper M, Yeager AM, Louie AC, Feldman EJ. Phase 2 trial of CPX-351, a fixed 5:1 molar ratio of cytarabine/daunorubicin, vs cytarabine/daunorubicin in older adults with untreated AML. Blood. 2014 May 22;123(21):3239-46. doi: 10.1182/blood-2013-12-540971. Epub 2014 Mar 31. PMID 24687088

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Started | 85 | 41
Completed | 36 | 18
Not Completed | 49 | 23

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin | Total
Number analyzed (Participants) | 85 | 41 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (4.63) | 68.2 (4.88) | 67.9 (4.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 16 | 48
  Male | 53 | 25 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission
Description: Response was defined according to International Working Group Criteria (Cheson, et al. 2003) which requires peripheral blood neutrophils of >1000/µL and peripheral blood platelets of >100,000/µL in the absence of bone marrow blasts.
Time Frame: Within 6 weeks of the last induction treatment
Population: Efficacy Evaluable Analysis Set: All randomized subjects who received at least 1 dose of study drug. One subject who developed Philadelphia chromosome positive disease prior to any efficacy assessment was excluded from the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
Participants | 41 | 20

2. Secondary Outcome: Remission Duration/Time to Remission
Description: Remission Duration was assessed from the time measurement criteria for CR were met until the first date that disease relapse was objectively documented or the subject died.
  Time to remission was measured from the date of randomization to the time measurement criteria for CR were first met.
Time Frame: Following achievement of CR over the study period
Population: Efficacy Evaluable Analysis Set
Measure: Median (Full Range); unit: days
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
days
  Remission Duration | 275 [40 to 730] | 235 [36 to 703]
  Time to Remission | 49 [32 to 163] | 40 [21 to 89]

3. Secondary Outcome: Event Free Survival
Description: Event-free survival begins from randomization to the date persistent disease is documented or date of relapse after CR, or death, whichever comes first.
Time Frame: Up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
days | 161 [116 to 226] | 55 [34 to 205]

4. Secondary Outcome: Overall Survival Rate at 1 Year
Description: Survival defined as the time from randomization to death.
Time Frame: 1 year
Population: Efficacy Evaluable Analysis Set
Measure: Number; unit: participants
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
participants | 39 | 18

5. Secondary Outcome: Rate of Stem Cell Transplant
Description: The rate of patients who underwent stem cell transplant.
Time Frame: Up to 1 year
Population: Efficacy Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
Participants | 13 | 10

6. Secondary Outcome: Aplasia Rate
Description: Bone marrow aplasia was defined as <20% cellularity and 5% blasts in the bone marrow aspiration evaluation.
Time Frame: Day 14 (1st Induction)
Population: Efficacy Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Number analyzed (Participants) | 84 | 41
Participants | 55 | 15

ADVERSE EVENTS:
Time Frame: Assessed during treatment period and recorded and reported any new serious adverse events (up to 30 days after completion of Treatment Period)
Description: The Safety Analysis Set included subjects receiving at least 1 dose of study drug and consisted of 126 subjects.
Arm/Group | Arm A: CPX-351 | Arm B: Cytarabine + Daunorubicin
Serious Adverse Events (participants affected / at risk) | 47/85 | 16/41
Other Adverse Events (participants affected / at risk) | 85/85 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: CPX-351 (N=85) | Arm B: Cytarabine + Daunorubicin (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Restrictive Cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 | 1
Ileal Perforation (Gastrointestinal disorders) | 1 | 0
Mouth Haemorrhage (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease Progression (General disorders) | 3 | 0
Infusion Related Reaction (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Graft Versus Host Disease (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 6 | 1
Catheter Site Cellulitis (Infections and infestations) | 1 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 0
Fungal Retinitis (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2
Pneumonia Fungal (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 7 | 2
Septic Shock (Infections and infestations) | 0 | 1
System Mycosis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Brain Herniation (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Nephrogenic Diabetes Insipidus (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 3 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Non-Cardiogenic Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: CPX-351 (N=85) | Arm B: Cytarabine + Daunorubicin (N=41)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 50 | 19
Neutropenia (Blood and lymphatic system disorders) | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 5
Angina Pectoris (Cardiac disorders) | 2 | 5
Atrial Fibrillation (Cardiac disorders) | 12 | 4
Bradycardia (Cardiac disorders) | 8 | 1
Tachycardia (Cardiac disorders) | 11 | 7
Conjunctivitis (Eye disorders) | 5 | 1
Abdominal Distension (Gastrointestinal disorders) | 11 | 6
Abdominal Pain (Gastrointestinal disorders) | 20 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 10 | 2
Ascites (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 43 | 23
Diarrhoea (Gastrointestinal disorders) | 56 | 27
Dry Mouth (Gastrointestinal disorders) | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 11 | 5
Dysphagia (Gastrointestinal disorders) | 6 | 2
Haemorrhoids (Gastrointestinal disorders) | 7 | 5
Mouth Haemorrhage (Gastrointestinal disorders) | 10 | 4
Mouth Ulceration (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 56 | 22
Oral Disorder (Gastrointestinal disorders) | 6 | 2
Oral Pain (Gastrointestinal disorders) | 6 | 0
Stomatitis (Gastrointestinal disorders) | 30 | 9
Toothache (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 23 | 12
Asthenia (General disorders) | 13 | 7
Catheter SIte Erythema (General disorders) | 17 | 6
Catheter Site Pain (General disorders) | 9 | 5
Chills (General disorders) | 33 | 13
Fatigue (General disorders) | 35 | 12
Gait Disturbance (General disorders) | 5 | 0
Oedema peripheral (General disorders) | 44 | 18
Oedema (General disorders) | 6 | 5
Pain (General disorders) | 9 | 3
Pyrexia (General disorders) | 26 | 14
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 | 3
Drug Hypersensitivity (Immune system disorders) | 5 | 1
Bacteraemia (Infections and infestations) | 10 | 2
Catheter Site Infection (Infections and infestations) | 5 | 5
Cellulitis (Infections and infestations) | 6 | 3
Clostridium difficile infection (Infections and infestations) | 9 | 0
Pneumonia (Infections and infestations) | 15 | 12
Transfusion Reaction (Injury, poisoning and procedural complications) | 10 | 2
Blood Alkaline Phosphate Increased (Investigations) | 5 | 0
Blood Creatinine Increased (Investigations) | 5 | 4
Breath Sounds Abnormal (Investigations) | 5 | 0
Cardiac Murmur (Investigations) | 8 | 1
Weight Decreased (Investigations) | 7 | 5
Weight Increased (Investigations) | 8 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 34 | 16
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Fluid Overload (Metabolism and nutrition disorders) | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Dizziness (Nervous system disorders) | 19 | 12
Dysgeusia (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 30 | 8
Lethargy (Nervous system disorders) | 6 | 0
Somnolence (Nervous system disorders) | 6 | 0
Syncope (Nervous system disorders) | 5 | 2
Tremor (Nervous system disorders) | 6 | 1
Anxiety (Psychiatric disorders) | 16 | 7
Confusional State (Psychiatric disorders) | 12 | 1
Depression (Psychiatric disorders) | 10 | 2
Hallucination (Psychiatric disorders) | 11 | 1
Insomnia (Psychiatric disorders) | 24 | 5
Mental Status Change (Psychiatric disorders) | 5 | 3
Haematuria (Renal and urinary disorders) | 5 | 2
Pollakiuria (Renal and urinary disorders) | 2 | 3
Renal Failure (Renal and urinary disorders) | 3 | 3
Renal Failure Acute (Renal and urinary disorders) | 5 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 5
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 1
Erythema (Skin and subcutaneous tissue disorders) | 10 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 8 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 28 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 6
Rash (Skin and subcutaneous tissue disorders) | 45 | 15
Skin Lesion (Skin and subcutaneous tissue disorders) | 6 | 1
Hypertension (Vascular disorders) | 16 | 6
Hypotension (Vascular disorders) | 15 | 10
Increased tendency to bruise (Blood and lymphatic system disorders) | 5 | 2
Gingival bleeding (Gastrointestinal disorders) | 3 | 3
Melaena (Gastrointestinal disorders) | 2 | 4
Proctalgia (Gastrointestinal disorders) | 6 | 0
Chest pain (General disorders) | 7 | 0
Bacterial disease carrier (Infections and infestations) | 5 | 2
Enterococcal bacteraemia (Infections and infestations) | 5 | 4
Staphylococcal bacteraemia (Infections and infestations) | 12 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 3
Purpura (Skin and subcutaneous tissue disorders) | 4 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 8 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No